CLINICAL TRIAL: NCT03739671
Title: Correlation of Vitamin D Supplementation in Emergency Medicine Residents and Seasonal Mood Symptoms
Brief Title: Vitamin D Supplementation and Effects on Mood in Emergency Medicine Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health South (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MMMC#1580
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Seasonal Mood Disorder
MeSH Terms: conditions — Seasonal Affective Disorder | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-vitamin D supplementation (Placebo Comparator): Group not receiving vitamin D supplementation
  Interventions: Dietary Supplement: No Vitamin D
- Vitamin D supplementation (Experimental): Group receiving vitamin D supplementation
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Group will receive 5000 units of vitamin D daily
  Arms: Vitamin D supplementation
Dietary Supplement: No Vitamin D — No vitamin D supplementation
  Arms: Non-vitamin D supplementation

SUMMARY:
Seasonal mood changes, and even feelings of depression, appear to have an association with decreased amounts of vitamin D in people living in geographic areas where exposure to sunlight during the winter months is relatively low. In this study, PGY-2 and PGY-3 Emergency Medicine residents at Lakeland Health will fill out PHQ-9 surveys for a total of 6 months (October-March), filled out at the end of each month. This is the time of year in southwest Michigan where exposure to direct sunlight is the lowest. The results of the individual surveys will be trended for the entire six months to see if individuals responds more positively after Vitamin D supplementation is initiated between months 3 and 4. Vitamin D supplementation will be 5000 units daily for the months of January-March.

ELIGIBILITY:
Inclusion Criteria:

* PGY-2 and PGY-3 Emergency Medicine Residents at Lakeland Health

Exclusion Criteria:

* Nonresidents and PGY-1 and PGY-4 Emergency Medicine residents at Lakeland Health

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Effect of vitamin D on resident mood | 6 months
  Using the Patient Health Questionnaire 9 (PHQ-9) survey results, data will be analyzed to determine if vitamin D helped increase positive responses as it correlates to mood. Using the Patient Health Questionnaire - 9 to determine the severity of the depressive moods. (Scaled from 0-27 with higher numbers being more severe. 0-4 is minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Lakeland Regional Healthcare, Saint Joseph, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided